CLINICAL TRIAL: NCT05028673
Title: Interventional, Randomized, Open-Label, Crossover, Single-Dose, Relative Bioavailability Study Comparing Two Pharmaceutical Formulations of Lu AG06466 and Investigating the Food Effect on Lu AG06466 in Healthy Subjects
Brief Title: A Study to Evaluate a New Tablet Formulation of Lu AG06466 in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: H. Lundbeck A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 19270A
Record Dates: First submitted 2021-08-25; First posted 2021-08-31 (Actual); Last update posted 2022-01-21 (Actual); Status verified 2022-01

CONDITIONS: Healthy
MeSH Terms: interventions — Antacids; aluminum hydroxide, magnesium hydroxide, drug combination

STUDY DESIGN:
Intervention Model Description: The first 3 periods will be randomized.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Lu AG06466 Capsule, Fasted State (Experimental): Participants will receive 1 capsule of Lu AG06466 in a fasted state.
  Interventions: Drug: Lu AG06466 Capsule
- Lu AG06466 Tablet, Fasted State (Experimental): Participants will receive 1 tablet of Lu AG06466 in a fasted state.
  Interventions: Drug: Lu AG06466 Tablet
- Lu AG06466 Tablet, Fed State (Experimental): Participants will receive 1 tablet of Lu AG06466 in a fed state (high-fat meal).
  Interventions: Drug: Lu AG06466 Tablet
- Lu AG06466 Tablet + Antacid, Fasted State (Experimental): Participants will receive 1 tablet of Lu AG06466 dosed in combination with antacid in a fasted state.
  Interventions: Drug: Lu AG06466 Tablet; Drug: Antacid

INTERVENTIONS:
Drug: Lu AG06466 Capsule — Hard capsule
  Arms: Lu AG06466 Capsule, Fasted State
Drug: Lu AG06466 Tablet — Film-coated tablet
  Arms: Lu AG06466 Tablet + Antacid, Fasted State; Lu AG06466 Tablet, Fasted State; Lu AG06466 Tablet, Fed State
Drug: Antacid — Oral suspension
  Other Names: Maalox; Aluminum hydroxide and magnesium hydroxide
  Arms: Lu AG06466 Tablet + Antacid, Fasted State

SUMMARY:
The main goal of this trial is to learn how a new tablet formulation of Lu AG06466 behaves in the body. Researchers will compare the new tablet formulation to the capsule formulation that is currently being tested in other clinical trials. They will measure the levels of the drug in the bloodstream for up to 3 days after participants take either the tablet or the capsule formulation. They will also look at whether the tablet formulation behaves differently when it is taken with and without food.

DETAILED DESCRIPTION:
This study will consist of 6 sequences with 4 periods (3 days/period) in each sequence. The first 3 periods will be randomized. Each Lu AG06466 dose administration will be separated by a washout period of at least 72 hours.

ELIGIBILITY:
Inclusion Criteria:

* The participant has a body mass index (BMI) ≥18.5 and ≤30 kg/m^2 at the Screening Visit and at the Baseline Visit.
* The participant is, in the opinion of the investigator, generally healthy based on medical history; a physical examination; vital signs; an electrocardiogram (ECG); and the results of the clinical chemistry, hematology, urinalysis, serology, and other laboratory tests at the Screening Visit and/or the Baseline Visit.

Exclusion Criteria:

* The participant has a personal history of a clinically significant psychiatric disorder (including severe affective disorder, severe anxiety disorder, psychotic tendencies, and drug-induced psychoses).
* The participant has or has had any clinically significant immunological, cardiovascular, respiratory, metabolic, renal, hepatic, gastrointestinal, endocrinological, hematological, dermatological, venereal, neurological, or psychiatric disease or other major disorder.

Other inclusion and exclusion criteria may apply.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2021-08-23 (Actual); Primary Completion 2021-12-29 (Actual); Study Completion 2021-12-29 (Actual)

PRIMARY OUTCOMES:
Area Under the Plasma Concentration-Time Curve From Time Zero to Infinity AUC(0-inf) of Lu AG06466 | 0 (predose) up to 72 hours postdose on Day 1 to Day 12
  AUC(0-inf) is defined as AUC0-tlast + Clast * t1/2 / ln2 (where Clast is the last quantifiable concentration and t1/2 is the apparent elimination half-life).
AUC(0-inf) of Metabolite Lu AG06988 | 0 (predose) up to 72 hours postdose on Day 1 to Day 12
  AUC(0-inf) is defined as AUC0-tlast + Clast * t1/2 / ln2 (where Clast is the last quantifiable concentration and t1/2 is the apparent elimination half-life).
Area Under Plasma Concentration-Time Curve from Zero to Last Quantifiable Concentration (AUC0-tlast) of Lu AG06466 | 0 (predose) up to 72 hours postdose on Day 1 to Day 12
AUC0-tlast of Metabolite Lu AG06988 | 0 (predose) up to 72 hours postdose on Day 1 to Day 12
Maximum Observed Plasma Concentration (Cmax) of Lu AG06466 | 0 (predose) up to 72 hours postdose on Day 1 to Day 12
Cmax of Metabolite Lu AG06988 | 0 (predose) up to 72 hours postdose on Day 1 to Day 12
Time to Reach Cmax (Tmax) of Lu AG06466 | 0 (predose) up to 72 hours postdose on Day 1 to Day 12
Tmax of Metabolite Lu AG06988 | 0 (predose) up to 72 hours postdose on Day 1 to Day 12
Apparent Oral Clearance (CL/F) of Lu AG06466 | 0 (predose) up to 72 hours postdose on Day 1 to Day 12
  CL/F is defined as dose / AUC0-inf.
Apparent Volume of Distribution (Vz/F) of Lu AG06466 | 0 (predose) up to 72 hours postdose on Day 1 to Day 12
  Vz/F is defined as CL/F * t1/2 / ln2.
Apparent Elimination Half-life (t1/2) of Lu AG06466 | 0 (predose) up to 72 hours postdose on Day 1 to Day 12
t1/2 of Metabolite Lu AG06988 | 0 (predose) up to 72 hours postdose on Day 1 to Day 12
Metabolic Ratio (MR) | 0 (predose) up to 72 hours postdose on Day 1 to Day 12
  MR is defined as AUC0-inf, Lu AG06988 / AUC0-inf, Lu AG06466.

CONTACTS AND LOCATIONS:
Locations (1):
- LabCorp Clinical Research Unit Ltd, Leeds, United Kingdom